CLINICAL TRIAL: NCT07229469
Title: Sumac Mouth Rinse in the Management of Recurrent Aphthous Stomatitis (A Randomized Controlled Clinical Study With Biochemical Assessment)
Brief Title: A Study on Sumac Mouth Rinse for Treating Recurrent Aphthous Stomatitis
Acronym: SUMAC-RAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-ReclM012315
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Aphthous Stomatitis
Keywords: Sumac, Rhus coriaria, mouth rinse, recurrent aphthous stomatitis, oral ulcers, TNF-alpha, anti-inflammatory, herbal therapy, clinical trial
MeSH Terms: conditions — Stomatitis, Aphthous; Oral Ulcer

STUDY DESIGN:
Intervention Model Description: A parallel, randomized controlled clinical trial with two groups: one group received Sumac mouth rinse and the control group received Tantum Verde mouth rinse . Participants were randomly assigned to each group. Both participants and the outcomes assessor were blinded to group allocation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and the outcomes assessor were blinded to the treatment allocation. The Sumac mouth rinse and placebo were identical in appearance, color, and packaging to maintain blinding throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Study group receiving sumac mouth rinse
  Interventions: Other: Sumac mouth rinse
- Control group (Active Comparator): Control group receiving tantum Verde mouth rinse
  Interventions: Drug: Tantum Verde mouth rinse

INTERVENTIONS:
Other: Sumac mouth rinse — Herbal mouth rinse containing Sumac extract
  Arms: Study group
Drug: Tantum Verde mouth rinse — Standard mouth rinse according to manufacturer instructions
  Arms: Control group

SUMMARY:
This randomized controlled clinical study aims to evaluate the effectiveness of a Sumac mouth rinse in the management of recurrent aphthous stomatitis (RAS). In addition to assessing clinical improvement in ulcer healing and pain reduction, biochemical analysis will be performed by measuring serum TNF-α levels to evaluate the anti-inflammatory effect of Sumac.

DETAILED DESCRIPTION:
Recurrent aphthous stomatitis (RAS) is one of the most common oral mucosal disorders, characterized by recurrent, painful ulcers that interfere with eating and speaking. The etiology of RAS is multifactorial and involves immune dysregulation and increased levels of inflammatory cytokines, particularly tumor necrosis factor-alpha (TNF-α).

Sumac (Rhus coriaria) is a natural herbal extract known for its anti-inflammatory, antioxidant, and antimicrobial properties. This randomized controlled clinical study aims to evaluate the clinical effectiveness of a Sumac mouth rinse in promoting ulcer healing and reducing pain among patients with recurrent aphthous stomatitis.

In addition to clinical assessment, biochemical evaluation of serum TNF-α levels will be performed before and after treatment to investigate the possible anti-inflammatory mechanism of Sumac. The study findings are expected to provide new insights into the potential therapeutic role of Sumac in managing RAS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Systemically healthy
* Patients with recurrent aphthous stomatitis minor type
* Duration of ulcer does not exceed 2 days
* Oral pain score of 4 or higher on the Visual Analog Scale (VAS)

Exclusion Criteria:

* Patients with poor oral hygiene
* Smokers and alcohol users
* Pregnant or lactating females
* Patients with a history of any topical or systemic medication or steroid therapy within 1 month prior to the study
* Vulnerable populations such as prisoners or individuals with mental or physical disabilities

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | At the baseline / Day 2 / Day 6
  Visual Analog Scale (VAS) to assess the intensity of oral ulcer pain reported by the patient, where 0 indicates no pain and 10 indicates the worst imaginable pain.
Ulcer size | At the baseline / Day 2 / Day 6
  Measurement of the oral ulcer diameter in millimeters using a ruler or photographic analysis to evaluate ulcer size reduction over time.

SECONDARY OUTCOMES:
Healing index | At the baseline / Day 2/ Day 6
  Healing index included four categories:
  1. Complete reepithelialization
  2. Incomplete reepithelialization
  3. Ulcer
  4. Tissue defect or necrosis
TNF- alpha | At the baseline/ Day 6
  Quantification of the inflammatory cytokine TNF-α in blood or saliva using ELISA to evaluate the inflammatory response associated with oral ulcers.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of oral medicine, Faculty of dentistry, Ain Shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided